CLINICAL TRIAL: NCT02533869
Title: The Optimization of a Low-dose Computed Tomography Protocol in Patients With Suspected Uncomplicated Acute Appendicitis (OPTICAP)
Brief Title: The Optimization of a Low-dose Computed Tomography Protocol in Patients With Suspected Uncomplicated Acute Appendicitis
Acronym: OPTICAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Paulina Salminen, MD, PhD, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPTICAP
Record Dates: First submitted 2015-08-18; First posted 2015-08-27 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Appendicitis; Other and Unspecified Acute Appendicitis; Acute Disease; Gastrointestinal Diseases; Intra-abdominal Infection
Keywords: low-dose computed tomography
MeSH Terms: conditions — Appendicitis; Acute Disease; Gastrointestinal Diseases; Intraabdominal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low-dose CT for acute appendicitis (Experimental): Low-dose computed tomography for diagnosing acute uncomplicated appendicitis Laparoscopic appendectomy
  Interventions: Radiation: Low-dose CT; Procedure: Laparoscopic appendectomy

INTERVENTIONS:
Radiation: Low-dose CT — Low-dose computed tomography for suspected acute uncomplicated appendicitis
Procedure: Laparoscopic appendectomy — All patients diagnosed with an uncomplicated acute appendicitis on low-dose CT-scan will undergo laparoscopic appendectomy to evaluate the sensitivity and specificity of the CT diagnosis

SUMMARY:
This study focuses on the use of contrast enhanced low-dose CT imaging as a modality to differentiate between uncomplicated and complicated acute appendicitis. Differentiation between the two forms of acute appendicitis is important because according to recent studies their treatment differs. Complicated forms are still treated operatively, while uncomplicated forms can be treated conservatively with antibiotics. In the initial phase of the study, several optimized CT protocols will be created with a phantom model. The two best performing models will be selected for the second phase of the study, in which patients presenting with suspected acute appendicitis will be imaged with the two protocols. All patients participating in the study will be treated operatively, primarily with a laparoscopic appendectomy. Thus histological confirmation for the diagnosis can be achieved and compared with the CT images. The goal of this study is to optimize a well-performing low-dose CT imaging protocol to use in the diagnosis of uncomplicated acute appendicitis.

DETAILED DESCRIPTION:
Acute appendicitis is one of the most common causes of abdominal pain in emergency departments as well as one of the most common indications for emergency abdominal surgery. The clinical diagnosis has been based on patient history, physical examination and laboratory findings as well as the "clinical eye" of the surgeon. Still the diagnosis remains challenging. One of the main problems is that many other disorders can mimic the clinical presentation of appendicitis, thus increasing the role of imaging techniques to aid in diagnostic accuracy. Now preoperative imaging in patients with suspected acute appendicitis is currently widely accepted as the standard of practice, and CT has been shown to clearly outperform US in terms of diagnostic performance. Nowadays, CT imaging is considered the primary imaging modality in the diagnosis for acute appendicitis as it is appraised for its high sensitivity and specificity. The main disadvantage of CT imaging is exposure to radiation. Thus the favorable diagnostic performance of CT imaging has encouraged optimization of protocols to minimize exposure to radiation through the development of low-dose CT protocols. Initial studies have indicated that contrast enhanced low-dose CT was not inferior to standard-dose contrast enhanced CT with no statistical significance in negative appendectomy rates, appendiceal perforation rates or patients requiring additional imaging.

This study focuses on the use of contrast enhanced low-dose CT imaging as a modality to differentiate between uncomplicated and complicated acute appendicitis. Differentiation between the two forms of acute appendicitis is important because according to recent studies their treatment differs. Complicated forms are still treated operatively, while uncomplicated forms can be treated conservatively with antibiotics. In the initial phase of the study, several optimized CT protocols will be created with a phantom model. The two best performing models will be selected for the second phase of the study, in which patients presenting with suspected acute appendicitis will be imaged with the two protocols. All patients participating in the study will be treated operatively, primarily with a laparoscopic appendectomy. Thus histological confirmation for the diagnosis can be achieved and compared with the CT images. The goal of this study is to optimize a well-performing low-dose CT imaging protocol to use in the diagnosis of uncomplicated acute appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Clinical suspicion of acute uncomplicated appendicitis based on history, physical examination, laboratory findings evaluated by a senior surgeon

Exclusion Criteria:

* Age <18 years or > 60 years
* Pregnancy or breastfeeding
* Allergy to contrast material or iodine
* History of appendectomy
* Renal failure, creatinine-value greater than the upper reference value
* Diabetes mellitus and metformin medication
* Suspicion of peritonitis and appendiceal perforation
* Incapability to cooperate and give consent to participate in the study
* A severe generalized disease or condition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
The specificity and sensitivity of low-dose CT in diagnosing acute uncomplicated appendicitis | Four months
  The sensitivity and specificity will be evaluated based on the operative and histopathological findings after laparoscopic appendectomy

SECONDARY OUTCOMES:
Negative appendectomy rate | Six months
Appendiceal perforation rate | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland